CLINICAL TRIAL: NCT04441983
Title: High-Resolution MRI (7 Tesla) Findings of the Plantar Plate Compared with Current Clinical Standard Sequences (1.5 or 3 Tesla) and Surgical Reference Standard
Brief Title: Foot/Ankle At 7T MRI
Status: Recruiting | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Reto Sutter, MD, head of radiology, medical doctor, principal investigator, Balgrist University Hospital
Other Study IDs: R449
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Plantar Plate Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: 7 Tesla MRI of the foot — 7 Tesla MRI

SUMMARY:
* To evaluate standard clinical sequences for 7 Tesla MRI of the foot and/or ankle to improve detailed depiction of the complex anatomy of this region.
* To evaluate various pathologies of the foot and/or ankle (plantar plate tears, Morton neuroma, tendon tears, ligament tears etc.).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* at least 18 years old
* Study group: Patients with specific pathologies (i.e. Morton neuroma, tendon tears, plantar plate tears) as proven by 1,5 or 3T MRI or asymptomatic subjects (to look at the normal microanatomy of different structures, mainly the plantar plate)
* Control group: No evidence of the respective pathology.

Exclusion Criteria:

* previous foot surgery with metal in vivo
* pregnancy or breast feeding
* any MRI contra-indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a forefoot MRI for clinical indications (or previous study) will be enrolled
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
sensitivity / specificity | 2 years
  The sensitivity/specificity for detection of various pathologies in the foot/ankle, for exampleMorton neuroma, plantar plate tears and tendon injuries at 7T MRI

CONTACTS AND LOCATIONS:
Overall Officials: Reto Sutter, MD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No